CLINICAL TRIAL: NCT07132684
Title: A Multicenter, Randomized, Controlled Clinical Trial Comparing VA and D/IA Induction Regimens in Elderly Patients With Acute Myeloid Leukemia Suitable for Intensive Chemotherapy
Brief Title: Comparison of VA and D/IA Induction Regimens in Elderly Fit Acute Myeloid Leukemia Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025095
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-07

CONDITIONS: AML, Adult
Keywords: acute myeloid leukemia; Older fit patients; venetoclax
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Daunorubicin; Idarubicin; Cytarabine; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D/IA (Daunorubicin/Idarubicin + Cytarabine) (Active Comparator): Induction Cycle 1:
  * Cytarabine: 100 mg/m²/day, days 1-7
  * Daunorubicin: 60 mg/m²/day, days 1-3 or
  * Idarubicin: 12 mg/m²/day, days 1-3
    • Induction Cycle 2 (if CR/CRi/CRh not achieved after Cycle 1):
  * Cyclophosphamide: 350 mg/m²/day, days 2 and 5o Cytarabine: 100 mg/m²/day, days 1-7
  * Daunorubicin: 45 mg/m²/day, days 1-2 or
  * Idarubicin: 8 mg/m²/day, days 1-2
  Consolidation Therapy
  • Intermediate-Dose Cytarabine (ID-Ara-C): 2 cycles Ara-C 1g/m² Q12h, d1-3 (aged ≥60 and <70 years) or Ara-C 500mg/m² Q12h d1-3 (aged ≥70 years)
  Maintenance Therapy
  * Low/Intermediate-Risk Patients:
    1. DA/IA "2+5" Regimen, 2 cycles Cytarabine: 100 mg/m²/day, days 1-5 Daunorubicin: 30 mg/m²/day, days 1-2 or Idarubicin: 8 mg/m²/day, days 1-2
    2. VA Regimen, 4 cycles Azacitidine: 75 mg/m²/day, days 1-5 Venetoclax: 400 mg/day, days 1-7, oral
  * High-Risk Patients:
  VA Regimen, 6 cycles
  Allogeneic Transplantation:
  Recommended for high-risk patients and those with persistent MRD positivity.
  Interventions: Drug: Daunorubicin/Idarubicin; Drug: Cytarabine; Drug: Azacitidine; Drug: Venetoclax
- VA Regimen (Experimental): Induction Cycles
  * Azacitidine: 75 mg/m²/day, days 1-7
  * Venetoclax:
  Day 1: 100 mg Day 2: 200 mg Days 3-21: 400 mg/day If bone marrow blasts >5% on day 21, extend to day 28 with 400 mg/day
  • Efficacy will be assessed after 2 cycles. If CR/CRi/CRh is not achieved but the investigator believes continued treatment is beneficial, up to 4 cycles may be administered.
  Consolidation Therapy • Intermediate-Dose Cytarabine (ID-Ara-C): 2 cycles Ara-C 1g/m² Q12h, d1-3 (aged ≥60 and <70 years) or Ara-C 500mg/m² Q12h d1-3 (aged ≥70 years)
  Maintenance Therapy
  * Low/Intermediate-Risk Patients:
    1: DA/IA "2+5" Regimen, 2 cycles Cytarabine: 100 mg/m²/day, days 1-5 Daunorubicin: 30 mg/m²/day, days 1-2 or Idarubicin: 8 mg/m²/day, days 1-2
    2.VA Regimen, 4 cycles Azacitidine: 75 mg/m²/day, days 1-5 Venetoclax: 400 mg/day, days 1-7, oral
  * High-Risk Patients:
    * VA Regimen, 6 cycles
  Allogeneic Transplantation:
  Recommended for high-risk patients and those with persistent MRD positivity.
  Interventions: Drug: Cytarabine; Drug: Azacitidine; Drug: Venetoclax

INTERVENTIONS:
Drug: Daunorubicin/Idarubicin — Daunorubicin/Idarubicin is used in Induction Therapy and Maintenance Therapy.
  Arms: D/IA (Daunorubicin/Idarubicin + Cytarabine)
Drug: Cytarabine — Cytarabine is used in Induction Therapy, Consolidation Therapy and Maintenance Therapy.
Drug: Azacitidine — Azacitidine is used in VA regimen
Drug: Venetoclax — Venetoclax is used in VA regimen

SUMMARY:
This study is a multicenter, randomized, controlled phase III clinical trial aimed at comparing the efficacy of two induction chemotherapy regimens-VA (Venetoclax + Azacitidine) and D/IA (Daunorubicin/Idarubicin + Cytarabine)-in elderly patients (aged 60-75) with acute myeloid leukemia (AML) who are fit for intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML according to WHO (2022) or ICC criteria.
* Age ≥60 and ≤75 years.
* ECOG performance status score of 0-2.
* Adequate organ function:

  * Total bilirubin ≤1.5× upper limit of normal (ULN)
  * AST and ALT ≤2.5× ULN
  * Serum creatinine <2× ULN
  * Cardiac enzymes <2× ULN
  * Left ventricular ejection fraction (LVEF, by echocardiogram) within normal range Signed informed consent by the patient or legal representative.

Exclusion Criteria:

* Acute promyelocytic leukemia with PML-RARA fusion gene.
* AML with RUNX1-RUNX1T1 or CBFB-MYH11 fusion genes.
* AML with BCR-ABL fusion gene.
* Relapsed or refractory AML (previously treated with induction chemotherapy, but hydroxyurea is allowed).
* Concurrent other malignancies requiring treatment.
* Active cardiac disease (e.g., uncontrolled angina, recent myocardial infarction, severe arrhythmias, uncontrolled heart failure, LVEF below normal).
* Severe infectious diseases (e.g., untreated tuberculosis, pulmonary aspergillosis).
* Other conditions deemed unsuitable by the investigator.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 1 years after completion of enrollment
  Time from randomization to death from any cause.

SECONDARY OUTCOMES:
Composite Complete Remission Rate (CR/CRh/CRi) | Six weeks after induction therapy
  Proportion of patients achieving CR, CRh, or CRi after induction.
MRD Negativity Rate | up to 1 years after completion of enrollment
  Proportion of patients achieving MRD negativity after induction and overall treatment.
Relapse-Free Survival (RFS) | up to 1 years after completion of enrollment
  Time from achieving CR/CRh/CRi to relapse or death.
Event-Free Survival (EFS) | up to 1 years after completion of enrollment
  Time from randomization to treatment failure, relapse, or death.
30-Day and 60-Day Mortality Rates | within 30 and 60 days of starting treatment.
  Proportion of patients who die within 30 and 60 days of starting treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wei, MD, Principal Investigator — Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Blood Diseases Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No